CLINICAL TRIAL: NCT02212015
Title: Single-arm, Multicenter, Open Label Phase II Trial to Evaluate the Efficacy of Pazopanib in Combination With Paclitaxel in Advanced and Relapsed Angiosarcoma
Brief Title: Evaluation of Votrient in Angiosarcoma
Acronym: EVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to interim analysis' results and definitions fixed in protocol
Sponsor: Heidelberg University (Other)
Collaborators: Universitätsmedizin Mannheim (Other); Helios Klinikum Berlin-Buch (Other); University Hospital Dresden (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Essen (Other); Hannover Medical School (Other); Klinikum der Universitaet Muenchen, Grosshadern (Other); Medical University of Vienna (Other); Medical University of Graz (Other); Medical University Innsbruck (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Peter Hohenberger, Prof. Dr. med., Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GISG-06
Record Dates: First submitted 2014-07-29; First posted 2014-08-08 (Estimated); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-01

CONDITIONS: Angiosarcoma
MeSH Terms: conditions — Hemangiosarcoma | interventions — pazopanib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib + Paclitaxel (Experimental): Paclitaxel administered every 28 days at day 1, day 8 and day 15 as a 2h intravenous infusion in a dose of 70mg/m2 in combination with pazopanib in a daily oral dose of 800mg (2x400mg)
  Interventions: Drug: Pazopanib + Paclitaxel

INTERVENTIONS:
Drug: Pazopanib + Paclitaxel — pazopanib in combination with paclitaxel in the treatment of patients with advanced or metastatic angiosarcoma.

SUMMARY:
Open-label phase II trial investigating the efficacy and safety of the investigational combination of pazopanib and paclitaxel.

DETAILED DESCRIPTION:
Open-label phase II trial investigating the efficacy and safety of the investigational combination of pazopanib and paclitaxel.This multi-center, open-label, prospective, single arm phase II study was designed to evaluate the clinical efficacy and safety of the experimental combination of pazopanib with paclitaxel in the treatment of patients with advanced or metastatic angiosarcoma.The safety evaluations (physical examination, laboratory checks as defined in protocol, toxicity/adverse event assessment according Eastern Cooperative Oncology Group version 4.0) are scheduled every cycle at day 1, 8, 15 and 29 (= day 1 of the next cycle).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments and must be willing to comply with treatment and follow-up. Note: Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging studies) and obtained prior to signing informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
* Age ≥ 18 years
* Life expectancy > 3 months
* Ability to swallow tablets
* Histological confirmed angiosarcoma, primary and secondary angiosarcoma (e.g. radiation-induced or angiosarcoma in chronical lymphedema) are eligible.
* Tumor must be locally advanced (unresectable) or metastatic. A progression must be documented within a 6-month period prior to screening.
* Eastern Cooperative Oncology Group performance status ≤ 2
* At least one measurable skin lesion or one measurable radiological (CT or MRI) target lesion (RECIST 1.1)
* Adequate organ system function as described in protocol
* A female is eligible to enter and participate in this study if she is either of non childbearing potential (defined in protocol) or childbearing potential with negative pregnancy test within 2 weeks prior to the first dose of study drug and agrees to use adequate contraception (as defined in protocol) during the study and for 30 days after the last dose of study drug.
* All sexually active male patients must agree to use adequate methods of birth control (see protocol) throughout the study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* Patients who need an active treatment for another malignant disease other than angiosarcoma
* Prior treatment with taxane within the last 12 months before study entry
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal sarcomatosis.(see protocol)
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding (see protocol)
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product (see protocol)
* Presence of uncontrolled infection
* QT prolongation interval (QTc) > 480 msec.
* Clinically significant cardiovascular disorders within the past 6 months
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer
* Poorly controlled hypertension (see protocol)
* Evidence of active bleeding or bleeding diathesis
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels
* Uncontrolled seizures, disorders of the CNS or psychiatric disorders which may put patient safety at risk, prevent giving informed consent or impact the patient's compliance with the use of study medication
* Women who are pregnant or breast feeding
* Patients who are not able or not willing to interrupt the intake of medications that are not allowed according to study protocol for at least 14 days before start of study medication and for the whole study period
* Chemotherapy or radiotherapy within 14 days before start of study medication
* Any ongoing toxicity from prior anti-cancer therapy that is > grade 1 and/or that is progressing in severity, except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2019-12-31 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hohenberger, MD, Principal Investigator — Universitätsmedizin Mannheim / Heidelberg University
Locations (10):
- Austria (2):
  - Universitätsklinik Graz, Graz
  - Universitätsklinik Wien, Vienna
- Germany (8):
  - Helios-Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Medical Center, Mannheim
  - Klinikum der Universität München Campus Großhadern, München

REFERENCES:
- See also: German Interdisciplinary Sarcoma Group — http://www.gisg.de
- See also: Sarcoma Platform Austria — http://www.sarcoma.at

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib + Paclitaxel: Paclitaxel administered every 28 days at day 1, day 8 and day 15 as a 2h intravenous infusion in a dose of 70mg/m2 in combination with pazopanib in a daily oral dose of 800mg (2x400mg) in the treatment of patients with advanced or metastatic angiosarcoma.
Period: Overall Study
Arm/Group | Pazopanib + Paclitaxel
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Subgroup 1 for Analyses [Count of Participants; unit: Participants] — Overall number of 26 participants were additionally subgrouped for outcome analyses (primary and secondary endpoint analyses) into cutaneous angiosarcomas versus visceral angiosarcomas
  Participants
    cutaneous angiosarcoma | 18
    visceral angiosarcoma | 8
Subgroup 2 for Analyses [Count of Participants; unit: Participants] — Overall number of 26 participants were additionally subgrouped for outcome analyses (primary and secondary endpoint analyses) into primary angiosarcomas versus secondary angiosarcomas
  Participants
    primary angiosarcoma | 13
    secondary angiosarcoma | 13

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression-free Survival
Description: The diagnosis of progession is based on tumor measurements assessed 182 days +/- 32 days after start of treatment (with imaging date as reference date) and according to the RECIST Version 1.1 criteria based on a predefined set of target lesions and non-target lesions.
Time Frame: 6 Month
Measure: Count of Participants; unit: Participants
Groups:
- Pazopanib + Paclitaxel: Paclitaxel i.v. infusion over 6 cycles, administered on day 1, day 8, day 15 of every cycle with a dosage of 70mg/m2 in combination with Pazopanib taken orally with a dosage of 800mg daily/once per day
  Pazopanib + Paclitaxel: pazopanib in combination with paclitaxel in the treatment of patients with advanced or metastatic angiosarcoma.
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Participants | 12
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Question is, if 6 months progression free survival rate (PFS-R) denoted by pPFS is higher than 35%. Test hypothesis is thus formulated as: H0: pPFS ≤0.35 versus H1: pPFS ≥0.35. This hypothesis is tested at the one-side significance level of 0.05. A 6 months PFS-R of 0.55 of cases or more is considered as clinically relevant success rate. The design is chosen such that rates of 0.55 or higher can be detected with a power of at least 0.8; Test type: Other; Rate = 0.46

2. Primary Outcome: Rate of Progression-free Survival, Subgroup 1 Analysis
Description: Rate of progression-free survival for Subgroup 1 categorizing the 12 participants who showed PFS after 6 months into cutaneous angiosarcoma versus visceral angiosarcoma The diagnosis of progession is based on tumor measurements assessed 182 days +/- 32 days after start of treatment (with imaging date as reference date) and according to the RECIST Version 1.1 criteria based on a predefined set of target lesions and non-target lesions.
Time Frame: 6 months
Population: Subgroup 1 (categorizing total number of 12 participants showing PFR survival after 6 months into cutaneous AS versus visceral AS)
Measure: Count of Participants; unit: Participants
Groups:
- Pazopanib + Paclitaxel: Paclitaxel i.v. infusion over 6 cycles, administered on day 1, day 8, day 15 of every cycle with a dosage of 70mg/m2 in combination with Pazopanib taken orally with a dosage of 800mg daily/once per day in the treatment of patients with advanced or metastatic angiosarcoma.
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 12
Participants
  cutaneous angiosarcoma | 11
  visceral angiosarcoma | 1
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Test type: Superiority; Rate difference = 0.486

3. Primary Outcome: Rate of Progression-free Survival, Subgroup 2 Analysis
Description: Rate of progression-free survival for Subgroup 1 categorizing the 12 participants who showed PFS after 6 months into primary angiosarcoma versus secondary angiosarcoma.
  The diagnosis of progession is based on tumor measurements assessed 182 days +/- 32 days after start of treatment (with imaging date as reference date) and according to the RECIST Version 1.1 criteria based on a predefined set of target lesions and non-target lesions.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 12
Participants
  primary angiosarcoma | 6
  secondary angiosarcoma | 6
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Test type: Superiority; Rate difference = 0

4. Secondary Outcome: Overall Survival
Description: Survival time of patient from start of treatment until death
Time Frame: from start of treatment until death within study's actual observation time for OS (22 months).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
months | 21.6 [20.5 to NA] — The upper bound of the 95% CI could not be estimated, because of too low number of events resulting in the curve representing the upper limit of confidence interval lying above 0.5.
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; The analysis of secondary endpoints is of descriptive nature and generally consists of summary statistics and interval estimation. Overall survival (OS) was defined as the time of start of treatment until death (event status=1) or last contact (censoring, event status=0). OS was analyzed using Kaplan-Meier curves. Median survival time is provided alonsgside two-sided 95% confidence interval (CI), if possible; Test type: Other; Median = 21.6

5. Secondary Outcome: Overall Survival, Subgroup 1 Analysis
Description: Survival time of patients from start of treatment until death, Subgroup 1 categorizing 26 overall participants into 18 cutaneous angiosarcoma versus 8 visceral angiosarcomas
Time Frame: from start of treatment until death within study's actual observation time for OS (22 months)
Population: Overall number of participants analyzed is 26. Thereof, 18 show cutaneous angiosarcoma, and 8 show cutaneos angiosarcoma.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
months
  cutaneous angiosarcoma: number analyzed (Participants) | 18
  cutaneous angiosarcoma | 21.6 [10.0 to 21.6]
  visceral angiosaroma: number analyzed (Participants) | 8
  visceral angiosaroma | 20.5 [2.8 to NA] — The upper bound of the 95% CI could not be estimated, because of too low number of events resulting in the curve representing the upper limit of confidence interval lying above 0.5.
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; The analysis of secondary endpoints is of descriptive nature and generally consists of summary statistics and interval estimation. Overall survival (OS) for subgroup 1 was defined as the time of start of treatment until death (event status=1) or last contact (censoring, event status=0). OS was analyzed using Kaplan-Meier curves. Median survival time is provided alonsgside two-sided 95% confidence interval (CI), if possible; Test type: Superiority; p = 0.752, Log Rank

6. Secondary Outcome: Overall Survival, Subgroup 2 Analysis
Description: Survival time of patients from start of treatment until death, Subgroup 2 categorizing 26 overall participants into 13 primary cutaneous angiosarcoma versus 13 secondary angiosarcomas
Time Frame: from start of treatment until death within study's actual observation time for OS (22 months)
Population: Overall number of participants analyzed is 26. Thereof, 13 show cutaneous angiosarcoma, and 13 show cutaneos angiosarcoma
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
months
  primary angiosarcoma: number analyzed (Participants) | 13
  primary angiosarcoma | 20.5 [10.0 to NA] — The upper bound of the 95% CI could not be estimated, because of too low number of events resulting in the curve representing the upper limit of confidence interval lying above 0.5.
  secondary angiosarcoma: number analyzed (Participants) | 13
  secondary angiosarcoma | 21.6 [NA to NA] — The upper and lower bound of the 95% CI could not be estimated, because of too low number of events resulting in curves representing the upper as well as the lower limit of confidence interval lying above 0.5.
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; The analysis of secondary endpoints is of descriptive nature and generally consists of summary statistics and interval estimation. Overall survival (OS) for subgroup 2 was defined as the time of start of treatment until death (event status=1) or last contact (censoring, event status=0). OS was analyzed using Kaplan-Meier curves. Median survival time is provided alonsgside two-sided 95% confidence interval (CI), if possible; Test type: Superiority; p = 0.621, Log Rank

7. Secondary Outcome: Response Rate (RR)
Description: Measurable skin lesions will be evaluated clinically and documented photographically, all other target lesions will be evaluated radiologically by CT or MRI according to RECIST Version 1.1.
  RR is given as 'Best overall response" BOR" defined as CR (complete remission), PR (partial) remission), SD (stable diesease) and PD (progressive disease) or NE (not evaluated) and provided by absolute and relative frequencies
Time Frame: determined every 8 weeks during first 6 month then every 12 weeks in follow-up period until progression or death or end of overall study observation period (22 months), then evaluated as BOR
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Participants
  CR | 2
  PR | 7
  SD | 6
  PD | 10
  NE | 1
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Test type: Other; Frequency of each category is given

8. Secondary Outcome: Response Rate (RR), Subgroup1 Analysis
Description: Measurable skin lesions will be evaluated clinically and documented photographically, all other target lesions will be evaluated radiologically by CT or MRI according to RECIST Version 1.1.
  RR is given as 'Best overall response" BOR" defined as CR (complete remission), PR (partial) remission), SD (stable diesease) and PD (progressive disease) or NE (not evaluated) and provided by absolute and relative frequencies for Subgroup 1 which is the analysis of cutaneous angiosarcoma versus visceral angiosarcoma
Time Frame: as for outcome 7
Population: Total number of participants analyzed is 26. Thereof, 18 show cutaneous AS, and 8 show visceral angiosarcoma
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Participants
  cutaneous angiosarcoma: number analyzed (Participants) | 18
  cutaneous angiosarcoma: CR | 2
  cutaneous angiosarcoma: PR | 6
  cutaneous angiosarcoma: SD | 4
  cutaneous angiosarcoma: PD | 6
  cutaneous angiosarcoma: NE | 0
  visceral angiosarcoma: number analyzed (Participants) | 8
  visceral angiosarcoma: CR | 0
  visceral angiosarcoma: PR | 1
  visceral angiosarcoma: SD | 2
  visceral angiosarcoma: PD | 4
  visceral angiosarcoma: NE | 1
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Response Rate (RR) is given as Best Overall Response (BOR) and given be absolute and relative frequencies. Categories of BOR are CR, PR, SD, PD and NE); Test type: Superiority; p = 0.349, Chi squared test, exact; Response Rate (RR) is given as Best Overall Response (BOR) and given be absolute and relative frequencies applied to the total of 26 enrolled subjects.. Categories of BOR are CR, PR, SD, PD and NE)

9. Secondary Outcome: Response Rate (RR), Subgroup 2 Analysis
Description: Measurable skin lesions will be evaluated clinically and documented photographically, all other target lesions will be evaluated radiologically by CT or MRI according to RECIST Version 1.1.
  RR is given as 'Best overall response" BOR" defined as CR (complete remission), PR (partial) remission), SD (stable diesease) and PD (progressive disease) or NE (not evaluated) and provided by absolute and relative frequencies for Subgroup 2 which is the analysis of primary angiosarcoma versus secondary angiosarcoma
Time Frame: as for outcome 7
Population: Total number of participants analyzed is 26. Thereof, 13 show primary angiosarcoma, and 13 show secondary angiosarcoma
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Participants
  primary angiosarcoma: number analyzed (Participants) | 13
  primary angiosarcoma: CR | 0
  primary angiosarcoma: PR | 5
  primary angiosarcoma: SD | 3
  primary angiosarcoma: PD | 5
  primary angiosarcoma: NE | 0
  secondary angiosarcoma: number analyzed (Participants) | 13
  secondary angiosarcoma: CR | 2
  secondary angiosarcoma: PR | 2
  secondary angiosarcoma: SD | 3
  secondary angiosarcoma: PD | 5
  secondary angiosarcoma: NE | 1
Statistical Analysis 1: Comparison: Pazopanib + Paclitaxel; Test type: Superiority; p = 0.385, Chi squared test, exact

10. Secondary Outcome: Adverse Events and Serious Adverse Events
Description: Number of patients in which adverse events occur during treatment according to Common Toxicity Criteria for Adverse Effects, Version 4.0
Time Frame: 30 days after EOS of last patient or end of overall study observation period (22 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Paclitaxel
Number analyzed (Participants) | 26
Participants
  Patients with AEs | 25
  Patients with SAEs | 10

ADVERSE EVENTS:
Time Frame: Adverse Events were collected over the study observation period which was 22 months
Groups:
- Pazopanib + Paclitaxel: Paclitaxel i.v. infusion over 6 cycles, administered on day 1, day 8, day 15 of every cycle with a dosage of 70mg/m2 in combination with Pazopanib taken orally with a dosage of 800 mg daily/once per day in the treatment of patients with advanced or metastatic angiosarcoma.
Arm/Group | Pazopanib + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib + Paclitaxel (N=26)
Lumbar spinal stenosis (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1)
Fever of unknown origin (General disorders) | 1 (1)
ALT increased (Hepatobiliary disorders) | 1 (1)
Reduced general condition (General disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Pain in thoracic spine (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilirubin increased (Hepatobiliary disorders) | 1 (1)
GOT increased (Hepatobiliary disorders) | 1 (1)
GPT increased (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib + Paclitaxel (N=26)
ALT increased (Hepatobiliary disorders) | 4 (12)
AST increased (Hepatobiliary disorders) | 4 (12)
Allergic reation to a drug (Product Issues) | 2 (2)
Reduced general condition (General disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9)
Anemia (Blood and lymphatic system disorders) | 3 (6)
Inappetance (Musculoskeletal and connective tissue disorders) | 4 (4)
Hypertension (Vascular disorders) | 12 (17)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Bilirubin increased (Hepatobiliary disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 16 (29)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 11 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Emesis (Gastrointestinal disorders) | 3 (8)
Acute nasopharyngitis (Infections and infestations) | 3 (3)
Erysipels (Infections and infestations) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Fever (General disorders) | 4 (4)
Pain foot (General disorders) | 4 (4)
Weight loss (Investigations) | 2 (2)
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 5 (11)
Tachycardia (Cardiac disorders) | 3 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Headache (Nervous system disorders) | 5 (6)
Leukopenia (Blood and lymphatic system disorders) | 6 (28)
Meteorism (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 12 (26)
Mucositis (General disorders) | 4 (6)
Nail dystrophia (Skin and subcutaneous tissue disorders) | 2 (3)
Neuropathia (Nervous system disorders) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 5 (18)
Obstipation (Gastrointestinal disorders) | 4 (7)
Dorsalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Vertigo (Nervous system disorders) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 6 (12)
Thoracical pain (General disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (14)
Oedema leg (General disorders) | 7 (11)
Exsikkosis (Metabolism and nutrition disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02212015/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02212015/SAP_001.pdf